CLINICAL TRIAL: NCT02365389
Title: Assiut University Hospital - Women Health Hospital
Brief Title: Once Daily In-situ Forming Versus Twice-daily Conventional Metronidazole Vaginal Gels for Treatment of Bacterial Vaginosis
Acronym: MNZ
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Omar Mamdouh Shaaban, Women Health hospital, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Vaginal gell
Record Dates: First submitted 2015-02-15; First posted 2015-02-18 (Estimated); Last update posted 2015-02-18 (Estimated); Status verified 2015-02

CONDITIONS: Vaginitis
MeSH Terms: conditions — Vaginitis

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Group A received in situ MTZ vaginal gel (Active Comparator): Received in situ MTZ vaginal gel once daily for 5 days. Treatment in this group was offered in the form of a bottle of an aqueous liquid (100 mL of a preparation composed of 0.8% MTZ, 20% pluronic F-127, 10% pluronic F-68, and 0.01% benzalkonium chloride). Women were asked to put 5 cc of the liquid into the vagina once daily for 5 days using a graded syringe and 10-cm long soft applicator.
  Interventions: Drug: MTZ vaginal gel
- Group B received conventional MTZ vaginal gel (Active Comparator): Group B (control group) received conventional MTZ vaginal gel (Tricho gel 0.8%, Sedico, Egypt) twice daily for 5 days, using the supplied nozzle, which applies about 5 gm of gel again in the same laying back position.
  Interventions: Drug: Conventional MTZ vaginal gel

INTERVENTIONS:
Drug: MTZ vaginal gel — MTZ vaginal gel once daily for 5 days
  Arms: Group A received in situ MTZ vaginal gel
Drug: Conventional MTZ vaginal gel — Conventional MTZ vaginal gel (Tricho gel 0.8%, Sedico, Egypt) twice daily for 5 days
  Arms: Group B received conventional MTZ vaginal gel

SUMMARY:
A previous study showed that in situ MTZ vaginal gel twice daily is more effective than the conventional vaginal gel product in sustained cure of BV( 4 weeks after treatment) (80.0% in the in-situ gel group as compared with 47.4 in the conventional gel group.The current study aims to compare the efficacy of the use of once daily in situ MTZ vaginal gel (0.8%) versus twice-daily conventional MTZ vaginal gel in treatment of BV.

DETAILED DESCRIPTION:
Bacterial vaginosis (BV) is one of the most frequently diagnosed infections in women attending genitourinary clinics. As 50% of cases of BV are asymptomatic, the true prevalence of this condition in the community is uncertain.Metronidazole (MTZ) is considered the drug of choice for the treatment of BV. It can be given either orally or locally. Formulations for the local administration of the drug include gels and suppositories.

The acceptance of suppositories is lower than the oral administration of the drug as they might cause irritation and thus affecting the patient's compliance. Moreover, the mode of administration of MTZ does not have a significant difference in the eradication of the pathogenic bacteria .

Among the metronidazole gels and lactic acid gels, for local application, lactic acid gels have been found to be more efficient and safer. The recurrence of BV is less common in patients treated with lactic acid gel when compared with patients treated with metronidazole gels. This may be attributed to the inhibition in the growth of the lactobacilli when MTZ is used for the treatment and depends on the concentration of the lactobacilli .

Intravaginal deliveries of MTZ for the treatment of BV have shown that there was an improvement in the clinical symptoms of the patients within 21-30 days of the starting of the treatment. Unfortunately, the vagina was not recolonized with lactobacilli within the stated period . The use of formulation consisting policarbophil-carbopol and lactic acid-chitosan mucoadhesive vaginal gels has also been reported and both of them have been found to be safe .

Cure rates following intravaginal treatment with MTZ account for 80-90% at the end of treatment and one month after the end of therapy. However, three months after the end of therapy the rate of relapses can overcome 30%. Persistence of an adherent bacterial biofilm, containing mostly Gardenerlla vaginalis is the main reason for failure of BV treatment .

Suppressive treatment with MTZ gel has been investigated with variable results . Moreover, long-term treatment with MTZ is not recommended because of the high incidence of gastrointestinal adverse reactions, the risk of peripheral neuropathy, and Candida super infection.

Although the patients are known to tolerate gels better than suppositories or ointments, the direct application of gels into the diseased sites of vagina might be difficult as well as improper. Therefore, vaginal therapy would be significantly improved if an intravaginally administered drug can retain at the site of administration for prolonged time .

The in situ forming hydrogel is a stimuli sensitive hydrogel that exists as an aqueous solution before administration. When exposed to external physical stimuli like heat, it undergoes reversible volume-phase transition, then immediately turned into standing gels after its contact with the mucosa .Recently, in situ gel drug delivery system has been investigated as a more convenient dosage form of topical applications. It's easy to be applied into the vagina with accurate dosing of liquid before turning to gel with even spreading. It had been tried before and proved effectiveness, safety and tolerance .

ELIGIBILITY:
Inclusion Criteria:

* Women with proven diagnosis of bacterial vaginosis infection from the Outpatient Gynecological Clinic in Women Health Center Assiut University.

Exclusion Criteria:

* Women refusal to participate in the study.
* Pregnant and nursing Women.
* Anticipation of difficulty of subsequent communication with the woman.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2014-05; Primary Completion 2014-10 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Clinical improvement of vaginitis. | 6 months
  Therapeutic success will be defined as the presence of at least 3 signs of Amsel's criteria (Milky, homogeneous, adherent discharge; vaginal pH > 4.5; release of fishy amine odor from vaginal fluid when mixed with 10% KOH (whiff test); and presence of > 20 of clue cells).